CLINICAL TRIAL: NCT02172417
Title: The Effect of Concomitant Cimetidine p.o. 400 mg t.i.d. and p.o. Ranitidine 300 mg Once Daily on Single Dose Pharmacokinetics of Tiotropium (14.4 µg) Given Intravenously Over 15 Minutes in Healthy Male and Female Subjects of 50-65 Years (Randomized, Open Label, Two Independent Two-fold Crossover)
Brief Title: Tiotropium in Combination With Concomitant Cimetidine or Ranitidine in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205.222
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Cimetidine; Tiotropium Bromide; Ranitidine

ARMS (2):
- Cimetidine + Tiotropium followed by Tiotropium (Experimental)
  Interventions: Drug: Cimetidine + Tiotropium; Drug: Tiotropium
- Ranitidine + Tiotropium followed by Tiotropium (Experimental)
  Interventions: Drug: Ranitidine + Tiotropium; Drug: Tiotropium

INTERVENTIONS:
Drug: Cimetidine + Tiotropium
  Arms: Cimetidine + Tiotropium followed by Tiotropium
Drug: Ranitidine + Tiotropium
  Arms: Ranitidine + Tiotropium followed by Tiotropium
Drug: Tiotropium

SUMMARY:
Study to investigate the effect of an inhibition of the renal cationic drug transporter on single dose pharmacokinetics of intravenous tiotropium in subjects in an age close to typical Chronic Obstructive Pulmonary Disease (COPD) population

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Age range from 50 to 65 years
* Within 20% of their normal weight (Broca index)

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, puls rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or with psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (≥ 24 hours) within ten half-lives of the respective drug before enrolment in the study or during the study (exclusion: ovarian hormone substitution)
* Use of any drugs which might influence the results of the trial within four weeks prior to administration or during the trial, among these all non-selective β-blockers, cromolyn sodium, nedocromil sodium, oral β-adrenergics or long-acting β-adrenergics such as salmeterol and formoterol, and anticholinergic drugs including ATROVENT® (ipratropium) by oral inhalation or ATROVENT® Nasal Spray
* Participation in another study with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 40 g/day)
* Drug abuse
* Blood donation (≥ 100 ml) within four weeks prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the reference range of clinical relevance
* Subjects with known hypersensitivity to anticholinergic drugs
* Subjects with known symptomatic prostatic hypertrophy or disturbed micturition
* Subjects with known narrow-angle glaucoma

In addition for female subjects (if appropriate):

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intra uterine pessary (IUP)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-07; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Cmax of plasma levels of tiotropium after dosing | up to 8 hours after i.v. treatment
Area under the curve (AUC) 0-4h of the plasma levels of tiotropium after dosing | 0 - 4 hours after i.v. treatment
Urinary excretion 0-4h after dosing (Ae0-4h) | 0 - 4 hours after i.v. treatment
Renal clearance of tiotropium (CLR) | pre-dose, 0-4 h, 4-8 h, 8-12 h, 12-24 , 24-28 h, 38-72 h and 72-96 h after i.v. treatment

SECONDARY OUTCOMES:
AUC 0-8h of plasma levels of tiotropium after dosing | 0-8 hours after treatment
Urinary excretion 0-96h after dosing (Ae0-96h) | 0-96 hours after treatment
Occurrence of Adverse Events | up to 4 - 8 days after last i.v. treatment
Changes from baseline in Laboratory Tests | Baseline, 4 - 8 days after last i.v. treatment
Changes in 12-lead electrocardiogram (ECG) | up to 24 h after i.v. treatment
Changes in Blood Pressure and Pulse Rate | up to 4 - 8 days after last i.v. treatment
Changes from baseline in physical examination | Baseline, 4 - 8 days after last i.v. treatment